CLINICAL TRIAL: NCT04169386
Title: A First-in-Human,Randomized, Double-Blind, Placebo-Controlled, Single Dose Escalation,Phase 1 Study to Evaluate the Safety,Tolerability, Pharmacokinetics and Pharmacodynamics of AK102 in Healthy Subjects
Brief Title: A Study of PCSK9 Inhibitor AK102 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: AD Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AK102-101
Record Dates: First submitted 2019-11-17; First posted 2019-11-19 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Hypercholesterolaemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- AK102 75mg (Experimental): AK102 75mg
  Interventions: Drug: AK102
- AK102 150mg (Experimental): AK102 150mg
  Interventions: Drug: AK102
- AK102 300mg (Experimental): AK102 300mg
  Interventions: Drug: AK102
- AK102 500mg (Experimental): AK102 500mg
  Interventions: Drug: AK102
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK102 — AK102 single dose administered subcutaneously
  Arms: AK102 150mg; AK102 300mg; AK102 500mg; AK102 75mg
Drug: Placebo — Placebo single dose administered subcutaneously
  Arms: Placebo

SUMMARY:
This is a first-in-human,randomized, double-blind, placebo-controlled, single dose escalation, phase 1 study to evaluate the safety, tolerability, PK/PD and immunogenicity of AK102 administered subcutaneously in healthy subjects. Subjects will be randomized into 4 planned single dose escalation cohorts or placebo cohort.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent.
* No clinically significant abnormalities judged by the principal investigator based on the medical history, physical examination, electrocardiogram and routine laboratory evaluations.
* Low-density lipoprotein cholesterol (LDL-C) level of 70-190 mg/dL (inclusive).
* Body mass index (BMI) ≥18 and ≤ 28 kg/m^2 , body weight >= 50 kg for male or >= 45 kg for female.

Exclusion Criteria:

* Triglyceride concentration >400 mg/dL (4.5 mmol/L).
* History of hypersensitivity reactions to any substance of the investigation drug or other monoclonal antibodies.
* Drug or alcohol abuse within 6 months prior to dosing.
* Blood pressure >140 mmHg (systolic) or > 90 mmHg (diastolic)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2018-11-22 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent AE | From single dose of AK102 through 12 weeks
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.

SECONDARY OUTCOMES:
Pharmacokinetic characteristics of AK102 | over 12 weeks
  Serum concentrations of AK102 at different timepoints before and after AK102 single dose.
Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) | At different time points from baseline through 12 weeks
  Low-Density Lipoprotein Cholesterol (LDL-C) blood concentrations before and after AK102 single dose.
Percent Change From Baseline in PCSK9 | At different time points from baseline through 12 weeks
  PCSK9 blood concentrations before and after AK102 single dose.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | At different time points from baseline through 12 weeks
  The immunogenicity of AK102 will be assessed by summarizing the number of subjects who develop detectable ADAs.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Chen, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No